CLINICAL TRIAL: NCT05137834
Title: The Effect of Postoperative Rehabilitation With a "Peanut Ball" After Total Knee Replacement. A Randomized Study Evaluating Postoperative Pain and Knee Function.
Brief Title: The Effect of Postoperative "Peanut Ball" Rehabilitation After Total Knee Replacement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02904
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with a "peanut ball". (Experimental): The rehabilitation program consists of mobility- and functional training exercises with a "peanut ball".
  Interventions: Other: Exercise
- Exercise without "peanut ball" (Active Comparator): The rehabilitation program consists of standard mobility- and functional training exercises without a "peanut ball".
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Post-surgical exercise

SUMMARY:
The purpose of this randomized controlled study is to evaluate the effect of postoperative exercise with a "peanut ball" after total knee replacement, on pain, intake of pain killers, knee function, and health-related quality of life.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be included in the study.

At baseline, before surgery, all patients will meet a nurse, a physical therapist, and an orthopedic doctor and answer questions about their health condition and do functional tests.

Each week is randomized to be either "peanut ball" or standard exercise week, with all patients during that week receiving the same treatment. Thus, depending on what week the patients are operated they will be mobilized with postoperative exercise with a "peanut ball" or to a standard exercise program (no peanut ball) 3-5 times/day for 6 weeks. All patients randomized to exercise with a "peanut ball" will receive a ball for free to bring home.

At the ward, the nurses will ask about the patient's pain level two times a day and register all medicines. The physical therapist will introduce the exercise and inform the patients to do the exercise 3-5 times/day a´ 15 minutes and fill in all exercises in an exercise diary.

2 weeks after surgery all patients have a standard visit to a nurse and a physical therapist at the orthopedic department. At this visit, the nurse will register the pain level and all intake of medicine and the physical therapist will measure the range of movement and the sit to stand test.

3 months after surgery all patients have a standard visit to a physical therapist at the orthopedic department. At this visit, all outcomes will be filled in or measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis planned for surgery with total knee replacement at Skåne University Hospital.

Exclusion Criteria:

* Patients who do not understand and talk the Swedish language
* Patients with dementia
* Revision surgery of the knee
* Unicompartmentmental knee replacement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) (0-100) | Change from baseline (before surgery) to 3 months after surgery
  The scale is from 0-100 and a higher value is associated with more pain. 0:no pain and 100: most possible pain.

SECONDARY OUTCOMES:
Range of movement | Change from baseline (before surgery) to 3 months after surgery
  The range of movement in the knee is measured with a goniometer. The range of movement may be between 0 degree to 145 degree. A higher degree is better.
Forgotten Joint Score (FJS) | Change from baseline (before surgery) to 3 months after surgery.
  Is a questionnaire of the patients awareness of their knee. Minimum score:0 (worse outcome), maximum score 100 (best outcome)
Knee injury and Osteoarthritis Outcome Score (KOOS-12) | Change from baseline (before surgery) to 3 months after surgery.
  Is a questionnaire of knee related function an quality of life. It consists of three parts: pain (4 items), function (4 items) and knee-specific quality of life (4 items). KOOS-12; in pain sub-item; In the sub-item of walking on a flat ground, going up and down stairs, sitting-reaching, function and daily life; There are patient-specific questions in the sub-item of quality of life, sitting up, standing, getting in and out of the car, turning the affected knee. The total scores obtained from the items in the KOOS-12 scale are calculated and the average of the total score is taken from the three sub-dimensions. If any of the three sub-item scores are missing, the average score cannot be calculated.
30 second sit to stand test | Change from baseline (before surgery) to 3 months after surgery.
  A test to evaluate leg strength and endurance. The 30 second stair stand asks participants to rise and sit back down in a chair as many times as they can during that time period, without using hands or arms for support. Higher scores mean better outcome (e.g. more stands in 30 seconds).
Euro Qol-five dimensions, Visual analogue scale (EQ-5D VAS) | Change from baseline (before surgery) to 3 months after surgery.
  Is a generic questionnaire about health related quality of life, 0-100, 0: The worst health you can imagine", 100: "the best health you can imagine". Patients are asked to indicate how your health is today and to write the number in an adoining box.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Skane, VO ortopedi, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No